CLINICAL TRIAL: NCT04240821
Title: Open-Label Extension Study of Theophylline for Treatment of Pseudohypoparathyroidism
Brief Title: Theophylline for Treatment of Pseudohypoparathyroidism
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Ashley Shoemaker (Other)
Responsible Party: Sponsor-Investigator, Ashley Shoemaker, Assistant Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 133013 Extension Study
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Pseudohypoparathyroidism; Pseudohypoparathyroidism Type 1a; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism

STUDY DESIGN:
Intervention Model Description: This is an open-label extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label theophylline (Experimental): Oral theophylline - either once daily capsule or q6h elixir.
  Interventions: Drug: Theophylline ER

INTERVENTIONS:
Drug: Theophylline ER — Oral theophylline
  Other Names: Theophylline elixir

SUMMARY:
Pseudohypoparathyroidism is a genetic disorder with limited treatment options, characterized by early-onset obesity, short stature, hormone resistance and cognitive impairment. This phase 2 clinical trial will test the efficacy of theophylline, a phosphodiesterase inhibitor, in pseudohypoparathyroidism. We hypothesize that theophylline will cause weight loss, improve glucose tolerance and decrease hormone resistance in children and young adults.

DETAILED DESCRIPTION:
Trial Objectives

1. The primary objective of this study is to evaluate the long-term safety of theophylline in patients with PHP.
2. The secondary objectives of this study are to evaluate changes in BMI, hormone resistance and epiphyseal closure associated with theophylline treatment of patients with PHP.

Study Design The proposed study is a single center, 24-month open label extension clinical trial for patients with PHP who complete the randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Successful completion of the randomized clinical trial "Phase 2 Study of Theophylline Treatment of Pseudohypoparathyroidism IND 133103 (11/1/2016)".

Exclusion Criteria:

1. History of a seizure disorder unrelated to hypocalcemia
2. History of a cardiac arrhythmia (not including bradycardia)
3. Hepatic insufficiency including cirrhosis and acute hepatitis (AST or ALT >3x upper limit of normal)
4. Congestive heart failure
5. Current cigarette use or alcohol abuse
6. Pregnancy or intention to become pregnant during the next year
7. Active peptic ulcer disease
8. Current use of medications known to effect theophylline levels
9. History of hypersensitivity to theophylline or other medication components
10. Unable to comply with study procedures in the opinion of the investigator

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 24 months
  Treatment-emergent adverse events will be compared before and during treatment

SECONDARY OUTCOMES:
BMI | 24 months
  Change in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: University faculty

REFERENCES:
- See also: Research Group Facebook Page — http://www.facebook.com/pseudohypoparathyroidism